CLINICAL TRIAL: NCT00397345
Title: Randomised,Double-blind,Placebo-controlled,Parallel Group Study TroVax, Added to First-line Standard of Care, Prolongs Survival of Patients With Locally Advanced or Metastatic Clear Cell Renal Adenocarcinoma.
Brief Title: TroVax Renal Immunotherapy Survival Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Oxford BioMedica (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TV3/001/06
Record Dates: First submitted 2006-11-08; First posted 2006-11-09 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Clear Cell Renal Carcinoma
Keywords: Renal; TroVax; survival; metastatic; Kidney; cancer; immunotherapy
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasm Metastasis; Neoplasms | interventions — TroVax

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Trovax (Experimental)
  Interventions: Biological: Trovax; Biological: Standard of care therapy
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo; Biological: Standard of care therapy

INTERVENTIONS:
Biological: Trovax — 1ml IM injection 2-8 weeks apart.
  Arms: Trovax
Biological: Placebo — Placebo
  Arms: Placebo
Biological: Standard of care therapy — subcutaneous low dose IL-2, interferon-α or sunitinib

SUMMARY:
The purpose of this study is to investigate whether TroVax, when added to first line standard of care therapy, improves survival for patients with locally advanced or metastatic clear cell renal adenocarcinoma.

DETAILED DESCRIPTION:
This is an international, randomised, double blind, placebo controlled, parallel group study to investigate whether a minimum of three doses of TroVax® added to first-line standard of care therapy, prolongs the survival of patients with locally advanced or metastatic renal clear cell adenocarcinoma.

The primary endpoint is survival. The study is designed to be pragmatic, limiting additional study related investigations to a minimum. Protocol mandated scans and X-rays are limited to two time points (baseline and week 26) to permit comparison of the percentage of patients with progressive disease at 6 months as a secondary efficacy endpoint. Six months was selected based on review of published literature indicating that progressive disease was commonly observed by 26 weeks in patients with renal cancer. Endpoints such as tumour response by RECIST are considered of secondary importance to survival and will be determined by radiological examinations ordered at the discretion of the investigator based on the clinical status of the patient and will be based the interpretation of the patient's care-team (investigator and local radiologist).

After signing the study informed consent form and meeting the baseline enrolment criteria patients will be assigned by the investigator (their physician) to one of the following defined first-line standard of care regimens based on what is best for the patient and consistent with local practice:

1. subcutaneous low dose IL-2
2. interferon-α (excluding pegylated IFNα)
3. sunitinib

TroVax® is administered at a dose of 1E9TCID50/ml in 1ml by injection into the deltoid muscle of the upper arm at regular intervals up to 8 weeks apart up to a maximum of 13 doses.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent. The patient must be competent to give written informed consent and comply with the protocol requirements.
* Locally advanced or metastatic, histologically proven clear cell renal carcinoma.
* Primary tumour surgically removed (some residual advanced primary tumour may remain).
* At least four weeks post surgery or radiotherapy.
* First-line. No prior therapy for renal cancer except surgery or radiotherapy.
* Measurable disease.
* Aged 18 years or more.
* Patient expected to survive a minimum of 12 weeks (i.e. in the opinion of the investigator there is a >90% probability that the patient will survive >12 weeks if treated with the selected standard of care).
* Free of clinically apparent autoimmune disease (including no prior confirmed diagnosis or treatment for autoimmune disease including Systemic Lupus Erythematosis, Grave's disease, Hashimoto's thyroiditis, multiple sclerosis, insulin dependant diabetes mellitus or systemic (non-joint) manifestations of rheumatoid disease).
* Total white cell count ≥ 3 x 109/L and lymphocyte count ≥1 x 109/L.
* Serum creatinine ≤1.5 times the upper limit of normal.
* Bilirubin ≤ 2 times the upper limit of normal and an SGPT of ≤ 4 times the upper limit of normal.
* Women must be either post menopausal, or rendered surgically sterile or, if of child bearing potential, must have been practising a reliable form of contraception (oral contraception + a barrier method) for at least three months prior to the first dose of TroVax® and must continue while they are being treated with TroVax®. Men must practise a reliable form of contraception (barrier or vasectomy) while they are being treated with TroVax®.
* No acute changes on 12-lead ECG.
* Ejection fraction documented as not less than 45% or no clinical suspicion that cardiac ejection fraction is less than 45%.(If clinical suspicion exists the ejection fraction should be measured according to local site procedures).
* Karnofsky performance status of ≥ 80%.

Exclusion Criteria:

* Cerebral metastases. (Known from previous investigations or clinically detectable).
* Previous exposure to TroVax®.
* Serious infections within the 28 days prior to entry to the trial.
* Known to test positive for HIV or hepatitis B or C.
* Life threatening illness unrelated to cancer.
* History of allergic response to previous vaccinia vaccinations.
* Known allergy to egg proteins.
* Known hypersensitivity to neomycin.
* Participation in any other clinical trial of a licensed or unlicensed drug within the previous 30 days or during the course of this trial.
* Previous malignancies within the last 10 years other than successfully treated squamous carcinoma of the skin or in situ carcinoma of the cervix treated with cone biopsy.
* Previous history of major psychiatric disorder requiring hospitalization or any current psychiatric disorder that would impede the patient's ability to provide informed consent or to comply with the protocol.
* Oral corticosteroid use unless prescribed as replacement therapy in the case of adrenal insufficiency.
* Ongoing use of agents listed in locally approved prescribing information as causing immunosuppression.
* Prior history of organ transplantation.
* Pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 733 (Actual)
Dates: Start 2006-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
overall survival | 18 months

CONTACTS AND LOCATIONS:
Locations (150):
- United States (45):
  - AZ Cancer Center, Tucson, Arizona
  - Little Rock Hematology / Oncology Associates, P.A., Little Rock, Arkansas
  - La Jolla, CA, La Jolla, California
  - The Angeles Clinic and Reseach Institute, Los Angeles, California
  - 1300 N. Vermont Ave, Los Angeles, California
  - UCLA Urology/Oncology, Los Angeles, California
  - Scripps Cancer Center, San Diego, California
  - Sharp Health Care, San Diego, California
  - UCHSC, Aurora, Colorado
  - Washington Cancer Center, Washington D.C., District of Columbia
  - Broward Oncology Associates, Fort Lauderdale, Florida
  - SCORE Physician Alliance, St. Petersburg, Florida
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Augusta Oncology Associates, Augusta, Georgia
  - SMO-USA Inc., Canton, Georgia
  - North Idaho Cancer Centre, Coeur d'Alene, Idaho
  - Patricia A. Joyce Cancer Institute, Olympia Fields, Illinois
  - Edward H Kaplan and Associates, Skokie, Illinois
  - St Francis Hospital, Indianapolis, Indiana
  - Cancer Care Centre of Indiana, New Albany, Indiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Henry Ford Health System / Josephine Ford Cancer Center, Detroit, Michigan
  - University Minnesota Fairview Medical Center, Minneapolis, Minnesota
  - Haematology and Oncology Associates at Bridgeport, Tupelo, Mississippi
  - Charleston Hematology and Oncology Associates,, Billings, Montana
  - Billings Clinical Research Center, Billings, Montana
  - Freedman Urology, Las Vegas, Nevada
  - Norris Cotton Cancer Center / Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - The Cancer Center @ HUMC, Hackensack, New Jersey
  - Columbia Presbyterian Medical Center, New York, New York
  - Pluta Cancer Centre, Rochester, New York
  - Piedmont Hospital, Inc., Canton, Ohio
  - Riverside Cancer Centre, Columbus, Ohio
  - Heamatology and Oncology Associates Inc., Columbus, Ohio
  - Flower Hospital/ Promedica Health System, Sylvania, Ohio
  - Oregon Urology Institute, Springfield, Oregon
  - Cancer Centre of the Carolinas, Greenville, South Carolina
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - University of Texas Medical Branch, Galveston, Texas
  - The Methodist Hospital, Houston, Texas
  - Urology Associates of South Texas, McAllen, Texas
  - Cancer Outreach Associates PC, Abingdon, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Madigan Army Medical Centre, Tacoma, Washington
- France (3):
  - CHU Besançon Hôpital Minjoz, Besançon
  - Centre Francois Baclesse, Caen
  - Centre François Baclesse-CLCC-Caen, Caen
- Universitätsklinikum C.G. Carus TU Dresden, Dresden, Germany
- Israel (6):
  - Oncology department, Assaf Harofeh Medical Center, Be’er Ya‘aqov, Zerifin
  - Oncology institute , Rambam /health Care Campus, Haifa
  - Meir Medical Center, Kfar Saba
  - Oncology department Rabin Medical center, Petah Tikva
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Oncology institute , The Chaim Sheba Medical center, Tel Litwinsky
- Poland (9):
  - IIndependent Public Hospital #1- , Oncology and Radiotherapy Dept, Gdansk
  - Holycross Oncology Center in Kielce, Department of Urology, Kielce
  - Maria Sklodowska-Curie Memorial Institute, Oncology Center Kraków Clinic Systemic and Generalized Neoplasms, Krakow
  - Independent Public Health Care Institution University Hospital in Krakow, Department of Oncology, Krakow
  - Lord's Transfiguration Independent Hospital Medical Academy Poznań, Poznan
  - Independent Public Clinical Hospital #2 - Pomeranian Medical Academy in Szczecin, Urology Clinic, Szczecin
  - Military Institute of Medicine, Department of Oncology, Warsaw
  - Maria Sklodowska-Curie Memorial Institute, Oncology Center in Warsaw, Clinic of Neoplasms of Urinary System, Warsaw
  - Regional Specialistic Hospital in Wrocław, Department of Urology, Wroclaw
- Romania (9):
  - Private Medical Centre, Arad
  - Fundeni Clinical Institute - Urology Department, Bucharest
  - Dinu Uromedica, Bucharest
  - "Prof. Dr. Th. Burghele" Clinical Hospital, Urology Clinic, Bucharest
  - "I. Chiricuta" Institute of Oncology, Cluj-Napoca
  - E-URO Medical Center, Cluj-Napoca
  - Provita Center SRL, Constanța
  - Sibiu Clinical County Hospital - Urology Clinic, Sibiu
  - Oncomed SRL, Timișoara
- Russia (40):
  - Leningrad Regional Oncological Center, Surgical Department #3, Saint Petersburg, Leningradskaya Oblast'
  - Republican Oncology Center" under the Ministry of Healthcare,, Petrozavodsk, Republic of Karelia
  - State Medical Institution of Healthcare: Clinical Oncological Center under the Ministry of Healthcare of the Republic of Tatarstan, Chemotherapy Department, Kazan', Tatarstan Republic
  - State Medical Institution: Arkhangelsk Regional Clinical Oncological Center, Surgery Department 7., Arkhangelsk
  - Chelyabinsk Regional Oncological Center, Chemotherapy Department, Chelyabinsk
  - State Therapeutical and Prophylactic Institution: Chelyabinsk Regional Oncological Center,, Chelyabinsk
  - Municipal Medical Institution: Oncological Center, Chemotherapy Department, Krasnodar
  - State Institution: Russian Oncological Research Center n.a. N.N. Blokhin of the Russian Academy of Medical Sciences, Department of Urology, Moscow
  - Russian Research Center of Roentgenology & Radiology , Surgery Department, Moscow
  - Russian State Medical University under the Federal Agency for Healthcare and Social Development, Department of Radiology Daignostics and Radiology Therapy, Moscow
  - Russian State Medical University under the Federal Agency for Healthcare and Social Development, Department of Urology and Surgical Nephrology, Moscow
  - Moscow Research Oncological Institute n.a. P.A. Hertzen, Urology Departmen, Moscow
  - Regional Research Clinical Institute n.a M.F. Vladimirskiy, Urology Department #1, Moscow
  - Non-State Medical Institution:Central Clinical Hospital, Moscow
  - Murmansk Regional Oncological Center, Oncology Department #5, Murmansk
  - Privolzhsky County Medical Center, Nizhny Novgorod
  - State Institution of Nizhny Novgorod Region: "Nizhny Novgorod Oncology Center", Department of Oncology #5 (for chemotherapy treatment), Nizhny Novgorod
  - Medical Radiological Research Center under the Russian Academy of Medical Sciences, Department of Urology, Obninsk
  - State Medical Institution: Omsk Regional Oncological Center, Chemotherapy Department, Omsk
  - Orenburg Regional Clinical Oncological Center, Chemotherapy Department, Orenburg
  - Regional State Medical Institution:"Orel Oncological Center", Oncology Department #5, Oryol
  - Pyatigorsk Branch of Stavropol Territorial Clinical Oncological Center (State Medical Institution), Outpatient Department, Pyatigorsk
  - Rostov State Medical University under the Federal Agency for Healthcare and Social Development, Department of Urology, Rostov-on-Don
  - Regional Clinical Oncological Center, Surgery Department, Ryazan
  - St. Petersburg State Pediatric Medical Academy, Saint Petersburg
  - Department of Urology, Saint Petersburg
  - Municipal Multi-Speciality Hospital #2, Department of Urology, Saint Petersburg
  - St. Petersburg State Medical Institution: Municipal Multi-Speciality Hospital #2, Department of Functional Diagnostics, Saint Petersburg
  - Municipal Hospital #26, Department Of Urology, Saint Petersburg
  - "Central Research Institute of Roentgenology & Radiology Federal Agency Healthcare Social Development", Saint Petersburg
  - Department of Biotherapy and Bone Marrow Transplantation, Saint Petersburg
  - St. Petersburg State Medical Institution: Municipal Hospital #15, Urology Department, Saint Petersburg
  - Samara Regional Oncology Center, Chemotherapy Department, Samara
  - "Oncological Center", Department of Haematology and Chemotherapy, Sochi
  - State Medical Institution: Stavropol Territorial Clinical Oncological Center, Department of Urology, Stavropol
  - State Medical Institution: Tambov Regional Oncological Center, Surgery Department, Tambov
  - State Higher Educational Institution: Siberian State Medical University, Department of Urology, Tomsk
  - Bashkir State Medical University, Urology Department, Ufa
  - State Medical Institution of Yaroslavl Region, Yaroslavl
  - State Institution of Mariy El Republic: "Republican Clinical Hospital", Department Of Urology, Yoshkar-Ola
- Spain (5):
  - Hospital Severo Ochoa, Servicio de Oncologia - Primera planta, Leganés, Madrid
  - Hospital de Cruces, Barakaldo
  - Hospital Santa Creu i Sant Pau Hospital Nuevo-Servicio de Oncologia Medica, Barcelona
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Marques de Valdecilla Consultas de Oncologia 1st planta, Santander
- Ukraine (17):
  - Bukovyna State Medical University, Department of Oncology, Radiodiagnostics and Radiotherapy, Chernivtsi
  - Dnepropetrovsk State Medical Academy, Department of Urology, Dnipro
  - Dnepropetrovsk State Medical Academy, Oncology, Radiodiagnostics and Radiotherapy Department, Dnipro
  - Donetsk Regional Antitumor Center, Urology Department, Donetsk
  - Ivano-Frankovsk State Medical University; Oncology Department, Ivano-Frankivsk
  - Kharkov Regional Clinical Urology and Nephrology Center, Oncourology Department, Kharkiv
  - Kharkov Medical Academy of Postgraduate Education, Oncology and Pediatric Oncology Department, Kharkiv
  - Urology Institute under the Ukrainian Academy of Medical Sciences, Oncourology Department, Kiev
  - Urology Institute under the Ukrainian Academy of Medical Sciences, Plastic and Reconstructive Urology Department, Kiev
  - Regional Public Institution: Krivoy Rog Oncological Center, Chemotherapy Department, Krivoi Rog
  - Lugansk Regional Clinical Oncological Center, Urology Department, Luhansk
  - Crimea State Medical University n.a. S.I. Georgievsky, Course in Urology at the Faculty Surgery#1 Department, Lviv
  - Odessa State Medical University;, Odesa
  - Crimean Republican Clinical Oncological Center, Chemotherapy Department, Simferopol
  - Uzhgorod National University,, Uzhhorod
  - Zaporozhye Medical Academy of Postgraduate Education, Oncology Department, Zaporizhzhya
  - Zaporozhye Medical Academy of Postgraduate Education, Urology Department, Zaporizhzhya
- United Kingdom (15):
  - Mount Vernon Cancer Centre, Northwood, Middlesex
  - Belfast City Hospital, Belfast, Northern Ireland
  - Clatterbridge Centre for Oncology, Bebington, Wirral
  - The Royal Bournemouth Hospital, Bournemouth
  - Bristol Haematology and Oncology Centre, Bristol
  - Beatson Oncology Centre, Glasgow
  - St Luke's Cancer Centre, Royal Surrey County Hospital, Guildford
  - St. James University Hospital, Leeds
  - Christie Hospital NHS Trust, Manchester
  - The James Cook University Hospital, Middlesbrough
  - University of Nottingham, Nottingham
  - The Churchill Hospital, Oxford
  - Weston Park Hospital, Sheffield
  - The South West Wales Cancer Institute, Swansea
  - New Cross Hospital, Wolverhampton

REFERENCES:
- [Result] Amato RJ, Hawkins RE, Kaufman HL, Thompson JA, Tomczak P, Szczylik C, McDonald M, Eastty S, Shingler WH, de Belin J, Goonewardena M, Naylor S, Harrop R. Vaccination of metastatic renal cancer patients with MVA-5T4: a randomized, double-blind, placebo-controlled phase III study. Clin Cancer Res. 2010 Nov 15;16(22):5539-47. doi: 10.1158/1078-0432.CCR-10-2082. Epub 2010 Sep 29. PMID 20881001